CLINICAL TRIAL: NCT03856385
Title: Impact of Mindful Walking Intervention on Daily Step Count: A Pilot Study
Brief Title: Impact of Mindful Walking Intervention on Daily Step Count
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Responsible Party: Principal Investigator, Heidi Zinzow, Associate Professor, Clemson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2017-099
Record Dates: First submitted 2019-02-12; First posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Walking (Experimental): Four weekly 60 minute sessions of mindful walking.
  Interventions: Behavioral: Mindful Walking
- Control (No Intervention): Weekly email messages encouraging physical activity.

INTERVENTIONS:
Behavioral: Mindful Walking — Weekly 60 minute mindful walking sessions involving observations of bodily sensations, experiences, and breath. Discussion of mindful walking experiences and encouragement to meet physical activity goals.
  Arms: Mindful Walking

SUMMARY:
Mindful walking is a meditation practice that combines physical activity and mindfulness practice. This study examined whether a mindful walking intervention increased physical activity and improved health outcomes. The investigators conducted a randomized experiment among adults with inadequate physical activity, whereby the intervention group received a four-week, one-hour-per-week mindful walking intervention and the control group received instructions to increase physical activity (N=38). Participants in both groups received a wrist-worn step count device as participation incentive. Physical activity and health outcomes were measured with an online survey and data obtained from the wearable device at baseline (T1), post-intervention (T2), and one month after the intervention (T3).

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18
* Able to read and understand English

Exclusion Criteria:

* Student athletes
* Medical condition that limits slow-paced walking for 20 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Rapid Assessment of Physical Activity Scale | one week
  self-report scale of physical activity, with total score ranging from 1-10; higher scores indicate increased activity
Daily Step Counts | one day
  Fitbit-HR device data
Screen Time | one week
  self-report measure, 4 items assessing television and non-television time in number of hours

SECONDARY OUTCOMES:
Perceived Stress Scale | one month
  self-report measure, total score ranges from 4 to 20, higher levels indicating higher levels of stress
Mental Health Inventory | one month
  self-report measure of health-related quality of life, total score ranging from 5 to 30, with higher levels indicating higher quality of life
Brief Edinburgh Depression Scale | 7 days
  self-report measure, total score ranging from 6 to 24, with higher levels indicating higher levels of depression symptoms
Freiburg Mindfulness Inventory | 7 days
  self-report measure, total score ranging from 14 to 56 with higher scores indicating higher levels of mindfulness skills
Pittsburgh Sleep Quality Index | one month
  self-report measure, total score ranging from 7 to 28, with higher scores indicating worse sleep quality

CONTACTS AND LOCATIONS:
Overall Officials: Lu Shi, Ph.D., Principal Investigator — Clemson University
Locations (1):
- Clemson University, Clemson, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared outside the research team